CLINICAL TRIAL: NCT00480623
Title: A Phase I Trial of Satraplatin Plus Radiation Therapy for Prostate Cancer Patients With Biochemical Recurrence Following Radical Prostatectomy
Brief Title: A Phase I Trial of Satraplatin Plus Radiation Therapy for Prostate Cancer Patients With Biochemical Recurrence
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT1-06-01
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Biochemical Failure; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — satraplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Satraplatin plus radiation therapy

SUMMARY:
This study is designed to measure the impact of Satraplatin plus radiation therapy to the bed of the prostate in patients who have developed biochemical failure of their prostate cancer. The main objective of this study is to determine the maximum tolerated dose and dose limiting toxicity for the combination of satraplatin and radiation therapy and to determine the recommended dose for subsequent Phase II trials.

DETAILED DESCRIPTION:
****Please Note: Dr.Howard Sandler's site will be open to accrual shortly, Dr. Sarantopoulos's site in San Antonio is open and recruiting patients.****

There were approximately 232,000 cases of prostate cancer diagnosed in the US in 2005. Most patients present with localized disease and undergo curative therapy, either radical prostatectomy (RP) or radiation therapy (RT). Although most men are cured after this therapy, approximately 30,000-50,000 annually in the US will develop recurrence after RP. For most of these patients, recurrence will be defined by biochemical recurrence (BCR), a rise in PSA with no other documented evidence of recurrence. Patients with BCR typically receive radiation therapy to the prostate bed. However, about 50% of these patients will develop distant recurrence outside of the pelvis and require systemic therapy.

Satraplatin is a third generation orally administered platinum compound. Early clinical studies demonstrated activity in tumors of the ovary and lung in addition to prostate cancer. Satraplatin has shown activity in prostate cancer in Phase II studies and has been evaluated in a pivotal Phase III study (The SPARC trial)as a single agent as second line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Over or equal to 18 years of age.
* ECOG performance status less than or equal to 1
* Adequate organ function.
* History of radical prostatectomy with histopathologic documentation of adenocarcinoma of the prostate.
* PSA over or equal to 0.2 ng/ml or less than or equal to 0.4 ng/ml. This includes patients whose PSA never becomes detectable. PSA progression must be measured by two consecutive samples, each separated by over or equal to 7 days. The PSA values of the two consecutive sample values must be greater than the previous (baseline) value, not greater than each other.

Exclusion Criteria:

* Known sites of measurable prostate cancer or bone scan positive for metastatic prostate cancer. (patients with a positive Prostascint scan will not be excluded)
* Prior therapy for prostate cancer except RP and neoadjuvant hormonal therapy. This includes chemo, hormonal (except neoadjuvant), RT, and biologic therapy.
* Lack of physical integrity of the upper GI tract, malabsorption syndromes, or inability to tolerate or absorb oral medications, including Crohn's disease and ulcerative colitis.
* Other concurrent immunotherapy, RT, chemotherapy,or ancillary therapy considered investigational (utilized for non-FDA approved indications and the context of a research investigation)and any chemotherapy not included in the study protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose and dose limiting toxicity for the combination of Satraplatin and radiation therapy. | Serum chemistry and CBC will be evaluated weekly. PSA level will be evaluated on Day on of week 5.

SECONDARY OUTCOMES:
PSA Response, Time to PSA Response, Duration of PSA response, Secondary Biochemical Recurrence Free Survival, Time to Biochemical Recurrence, Effect of Satraplatin on Serum Testosterone Levels, Safety and Tolerability. | PSA level will be evaluated on Day on of week 5. There will be an end of treatment visit within 30 days of the last RT-Satraplatin treatment. PSA will be drawn every 3 m for 2 years, then every 6 m until evidence of either PSA or clinical progression.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Sandler, MD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin